CLINICAL TRIAL: NCT06269263
Title: Pilot Study to Determine Feasibility of Home-based Cardiac Rehabilitation in Patients With Chronic Heart Failure (Pilot-CRHF)
Brief Title: Feasibility of Home-based Cardiac Rehabilitation in Patients With Chronic Heart Failure (Pilot-CRHF)
Acronym: Pilot-CRHF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 339/23-ek
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Pilot study of home-based cardiac rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based cardiac rehabilitation (Experimental): Home-based cardiac rehabilitation
  Interventions: Behavioral: Home-based cardiac rehabilitation

INTERVENTIONS:
Behavioral: Home-based cardiac rehabilitation — Guided by physiotherapists, patients will receive different trainings regrading endurance/balance/resistance,/coordination at home

SUMMARY:
The proposed study will determine the willingness of patients for participation. Furthermore, the assessment of tests to identify eligible patients and the type of exercise intervention that goes along with a high patient compliance is crucial. Also, more information about possible factors preventing patients from participating is required. Therefore, if the patient is willing to participate, the investigators will assess patients' medical history, medication and QoL as well as parameters of routine diagnostics (i.e. echocardiography, laboratory testing, MRI). Following, while the in-patient stay due to cardiac decompensation, the investigators will conduct several assessment-tests to determine the physical status, the exercise capacity and the cognitive function. Moreover, physiotherapists will instruct the patients in the exercise program. After discharge from the hospital, physiotherapist will visit the patient at home to instruct them again in the exercises. Then, the patients will conduct the program on their own for a period of 12 weeks. During the exercise period, a doctoral student will visit the patients at home every 3 weeks to check whether they are doing the exercises correctly and to determine whether there are any problems with the program. After the exercise period of 12 weeks, the baseline characteristics will be assessed again at the University Hospital Leipzig.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure irrespective of the ejection fraction
* Recent history of acute cardiac decompensation leading to hospitalization

Exclusion Criteria:

* Patients not willing to participate
* Patients with orthopedic diseases limiting their mobility
* Cognitive diseases that hinder adequate participation in the opinion of the investigator
* Inpatient rehabilitation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing the program | After 12 weeks
  Percentage of patients completing the program

SECONDARY OUTCOMES:
Quality of life by KCCQ | After 12 weeks
  QoL measured by Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ measures in values from 0 to 100 with higher values indicating better quality of life
Exercise capacity | After 12 weeks
  Exercise capacity measured by 6-minutes walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of main study results
Access Criteria: Upon reasonable request by other researchers